CLINICAL TRIAL: NCT03231644
Title: Fibrous Dysplasia, McCune-Albright Syndrome Patient Registry
Status: Recruiting | Type: Observational
Sponsor: Tovah Burstein (Other)
Responsible Party: Sponsor-Investigator, Tovah Burstein, Community Engagement Director, Fibrous Dysplasia Foundation
Organization: Fibrous Dysplasia Foundation (Other)
Other Study IDs: Pro00018980.
Record Dates: First submitted 2017-07-20; First posted 2017-07-27 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Fibrous Dysplasia; McCune Albright Syndrome; Mazabraud Syndrome
Keywords: Fibrous Dysplasia; McCune-Albright Syndrome; Mazabrauds; FD/MAS
MeSH Terms: conditions — Fibrous Dysplasia of Bone; Fibrous Dysplasia, Polyostotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- FD/MAS Patients: Patients with fibrous dysplasia and/or McCune-Albright syndrome and related disorders.

SUMMARY:
The FD/MAS Patient Registry is an IRB-approved research study that that invites the patients and families to help answer some of the biggest questions about FD/MAS by completing questionnaires about their lives with FD or MAS.

Have you enrolled in the FD/MAS Patient Registry yet? Are you up-to-date on your surveys? Take a trip to www.fdmasregistry.org today to learn more about the project, enroll, complete your surveys, or make sure you aren't due to provide more info!

The FD/MAS Patient Registry: Your story powers research.

DETAILED DESCRIPTION:
The FD/MAS Patient Registry is an IRB approved research project that allows patients and families to share their experiences with fibrous dysplasia/McCune-Albright syndrome (FD/MAS) by completing a series of surveys.

The surveys were created in collaboration with patients, parents, clinicians and researchers, so that the data can be used to answer some of the most important questions about FD/MAS, including:

the way the disease develops over time (its "natural history"), the patient experience of the disease, and its impact on quality of life, how and when diagnoses are made, the scope of treatments in use, what surgical techniques work best, and for whom, what other medical interventions work best, and for whom, what social services and therapies are useful, the costs of care to patients and their families, issues that concern patients (such as the impact of pregnancy on FD, or children feeling different and facing stigma), and which research questions and support programs you think are important to fund.

Participation is free and convenient for people with FD/MAS and their legal guardians. You can join today at www.fdmasregistry.org.

ELIGIBILITY:
Inclusion Criteria any one or more of the following:

* clinical diagnosis of fibrous dysplasia
* clinical diagnosis of McCune-Albright syndrome
* clinical diagnosis of Mazabraud's syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community sample of all patients in these particular disease communities.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-10-31 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Treatment satisfaction | Through study completion, an average of every 2 years
  FACIT-Treatment Satisfaction scale
Perceived symptoms of pain | Through study completion, an average of every 2 years
  Brief Pain Inventory
Depression/anxiety | Through study completion, an average of every 2 years
  Hospital Anxiety Depression Scale
Stigma | Through study completion, an average of every 2 years
  NeuroQol Pediatric and Adult Stigma short forms
Health-related Quality of Life | Through study completion, an average of every 2 years
  SF-36,PedsQL 4.0
Financial health | Through study completion, an average of every 2 years
  FACIT-Cost

CONTACTS AND LOCATIONS:
Locations (1):
- Tovah Burstein, Bethesda, Maryland, United States